CLINICAL TRIAL: NCT07363460
Title: A Randomized, Double-blind, Placebo-controlled Phase II Clinical Trial to Evaluate the Efficacy and Safety of HSK39297 Tablets in Patients With Lupus Nephritis
Brief Title: Study to Assess Efficacy and Safety of HSK39297 Tablets in Patients With LN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK39297-205
Record Dates: First submitted 2025-12-03; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Lupus Nephritis (LN)
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 200mg QD (Active Comparator): Patients take double-blind HSK39297 tablets 200mg for 52 weeks
  Interventions: Drug: HSK39297 200mgQD
- 300mg QD (Active Comparator): Patients take double-blind HSK39297 tablets 300mg for 52 weeks
  Interventions: Drug: HSK39297 300mgQD
- Placebo (Placebo Comparator): Patients take double-blind placebo for 52 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSK39297 200mgQD — once daily, oral administration of HSK39297 tablets 200mg from Day 1 to Week 52.
  Arms: 200mg QD
Drug: HSK39297 300mgQD — once daily, oral administration of HSK39297 tablets 300mg from Day 1 to Week 52.
  Arms: 300mg QD
Drug: Placebo — once daily, oral administration of placebo from Day 1 to Week 52.
  Arms: Placebo

SUMMARY:
A double-blind,placebo controlled,randomized Phase 2 study to evaluate the safety and tolerability of once-daily, oral administration of 200 or 300 mg HSK39297 tablets versus placebo in Patients With Lupus Nephritis

ELIGIBILITY:
Inclusion Criteria:

1. Understand and comply with the research requirements, voluntarily participate in the research and sign the informed consent form before starting the relevant procedures;
2. Age ≥ 18 and < 75 years old at screening, gender not limited;
3. Positive anti-ANA antibody and/or anti-dsDNA antibody (research center);
4. Pathological type of active III or IV lupus nephritis confirmed by renal biopsy within 12 months before screening, with or without type V (adopting the 2003 International Society of Nephrology/Renal Pathology Working Group's lupus nephritis pathological classification criteria, see Appendix 2; for recurrent subjects, the investigator assesses whether a repeat renal biopsy is necessary; renal biopsy is conducted after confirming that the subject meets all other inclusion criterias and does not meet the exclusion criterias);
5. Evidence of active lupus nephritis exists, and the investigator assesses that it is necessary to receive glucocorticoid combined with MMF treatment. Active lupus nephritis must meet the following two criterias:

   a) Proteinuria:

   a) At screening: 24h-UPCR ≥ 1g/g or FMV-UPCR ≥ 1g/g or FMV-UACR ≥ 0.5g/g; b) Before randomization: 24h-UPCR ≥ 1g/g (central laboratory); b) At screening: SLEDAI-2000 ≥ 8;
6. First onset or recurrence of lupus nephritis (for subjects who have received MMF treatment previously and have experienced recurrence, the investigator and the sponsor jointly assess the benefit based on the study's medication regimen to determine whether they can be enrolled);
7. Female subjects with reproductive capacity [excluding those who have undergone surgical sterilization (hysterectomy, bilateral tubal ligation, bilateral oophorectomy) at least 6 weeks prior to screening or who are postmenopausal (defined as having no menstruation for 12 months, with no other medical cause)]; a negative pregnancy test must be confirmed during the screening period. The subject must agree not to attempt pregnancy and not to donate oocytes from the date of signing the informed consent form until at least 30 days after the last administration of investigational product, and must use effective contraception; male subjects must agree not to donate sperm for at least 90 days from the date of signing the informed consent form until at least 90 days after the last administration of investigational product, and must use highly effective contraception with their female partners (see Appendix 3).

Exclusion Criteria:

1. The subject has previously failed to respond to treatment with MMF or other mofetil mycophenolate drugs, as assessed by the investigator.
2. Allergy to the investigational product or MMF, or contraindications to MMF and glucocorticoids.
3. Currently receiving or requiring administration of any drug listed in Section 5.7.2.2 "Prohibited Concomitant Medications" during the study period.
4. Receiving systemic glucocorticoid therapy for reasons other than systemic lupus erythematosus or lupus nephritis at screening (dose > 10 mg/day prednisone or equivalent; dosage conversion details see Appendix 4).
5. Received treatment with other investigational drugs within 30 days prior to screening or within 5 half-lives (whichever is longer).
6. Presence of rapidly progressive glomerulonephritis at screening (eGFR decline exceeding 50% within 3 months, or less than 50% but with rapid decline risk assessed by the investigator); renal biopsy showing crescents occupying more than 50% of glomeruli, or glomerulosclerosis exceeding 60%, or tubular atrophy/interstitial fibrosis exceeding 60%.
7. Presence of severe extra-renal manifestations of systemic lupus erythematosus at screening, including but not limited to severe pulmonary hypertension (WHO classification IV or higher), severe pulmonary interstitial fibrosis, severe myocarditis, severe heart failure (NYHA classification IV), or active central nervous system lupus.
8. Major, unstable, or uncontrolled acute or chronic diseases affecting various systems (e.g., cardiovascular, respiratory, hematological, gastrointestinal, hepatic, renal, neurological systems) within 6 months prior to screening or at screening that may affect study results or place the subject at high risk, excluding those caused by SLE.
9. History of other autoimmune diseases.
10. History of any of the following infections:

1) History of encapsulated bacterial infection (e.g., Neisseria meningitidis, Streptococcus pneumoniae, Haemophilus influenzae) within 1 year prior to screening; 2) Active tuberculosis at screening; history of active tuberculosis within 2 years prior to screening; history of active tuberculosis currently cured but assessed by the investigator to be at risk for reactivation; positive interferon-gamma release assay with determination by the investigator or consulting specialist physician that it represents latent tuberculosis requiring prophylactic anti-tuberculosis treatment; 3) History of other active infections requiring antimicrobial treatment within 3 months prior to screening.

11. History of major organ (heart, lung, kidney, liver) transplantation or hematopoietic stem cell/bone marrow transplantation, or planned for transplantation.

12. Currently undergoing regular hemodialysis or planning to undergo hemodialysis during the study period.

13. History of gastrointestinal surgery that may significantly affect drug absorption, distribution, metabolism, and excretion, or history of severe gastrointestinal disease, or difficulty in swallowing, frequent vomiting leading to difficulty in eating or taking medication.

14. Diagnosis of malignancy within 5 years prior to screening, excluding basal cell carcinoma of the skin, papillary thyroid carcinoma, squamous cell carcinoma of the skin, or cervical carcinoma in situ.

15. Major surgical procedures within 6 months prior to screening. 16. Laboratory tests at screening meet any of the following criteria:

1. Estimated Glomerular Filtration Rate (eGFR) < 30 ml/min/1.73m² (calculated by CKD-EPI 2021 formula, see Appendix 5);
2. Hematology: neutrophils < 1 × 10⁹/L; leukocytes < 2 × 10⁹/L; hemoglobin < 80 g/L; platelets < 50 × 10⁹/L;
3. Liver function: Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) ≥ 3 × ULN; Total Bilirubin (TBIL) ≥ 2 × ULN;
4. Hepatitis B virus surface antigen (HBsAg) positive, or HBsAg negative but Hepatitis B virus core antibody (HBc-Ab) positive with HBV-DNA detection result higher than the quantitative lower limit; Hepatitis C virus antibody (HCV-Ab) positive;
5. Human Immunodeficiency Virus antibody (HIV-Ab) positive. 17. Pregnant or lactating female subjects at screening. 18. Other situations deemed unsuitable for participation by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2027-11-05 (Estimated); Study Completion 2028-07-06 (Estimated)

PRIMARY OUTCOMES:
Ratio of 24h-UPCR compared to Baseline | 24 weeks
  Urine Protein Creatinine Ratio

SECONDARY OUTCOMES:
Proportion achieving CRR/PRR | 12,24,52 weeks
  Complete Renal Response,Partial Renal Response
Proportion achieving CRR/PRR without renal recurrence | 24,52 weeks
  Complete Renal Response,Partial Renal Response
Proportion achieving CRR/PRR with glucocorticoid ≤ 5mg/d | 24,52weeks
  Complete Renal Response,Partial Renal Response
Proportion achieving 25%/50% reduction in 24h-UPCR | 12,24,52 weeks
  Urine Protein Creatinine Ratio
Time to first achievement of CRR, 25%/50% proteinuria reduction | from baseline to 52 weeks
  Complete Renal Response
Duration of sustained CRR/PRR | from baseline to 52 weeks
  Complete Renal Response,Partial Renal Response
Change in 24h-UPCR from baseline. | from baseline to 52 weeks
  Urine Protein Creatinine Ratio
Change in eGFR from baseline | 12,24,52 weeks
  Estimated glomerular filtration rate
Proportion with Glucocorticoid dose ≤ 5mg/d | 24,52 weeks
Annualized slope of eGFR | 52 weeks
  Estimated glomerular filtration rate
Change in SLEDAI-2000 (Systemic lupus erythematosus disease activity index 2000，SLEDAI-2000)total score from baseline | 12, 24, 52 weeks
  SLEDAI-2000 scale ranges form 0 to 105 score. The higher scores indicate a higher disease activity level of the subject's systemic lupus erythematosus .
Incidence and severity of adverse events (AEs) | 52 weeks
Pharmacokinetic characteristics(Cmax) of HSK39297 tablets in plasma. | 52 weeks
Pharmacokinetic characteristics(Cmin) of HSK39297 tablets in plasma. | 52 weeks
Pharmacokinetic characteristics(Cavg) of HSK39297 tablets in plasma. | 52 weeks
Pharmacokinetic characteristics(Tmax) of HSK39297 tablets in plasma. | 52 weeks
Pharmacokinetic characteristics(AUC0-τ) of HSK39297 tablets in plasma. | 52 weeks
Changes from baseline of pharmacodynamic indicators(Ap) | 52 weeks
Changes from baseline of pharmacodynamic indicators(Bb) | 52 weeks
Changes from baseline of pharmacodynamic indicators(sC5b-9) | 52 weeks
Changes from baseline in biological markers （C3）reflecting immunological activity of lupus nephritis | 52 weeks
Changes from baseline in biological markers （C4）reflecting immunological activity of lupus nephritis | 52 weeks
Changes from baseline in biological markers （anti-dsDNA antibody）reflecting immunological activity of lupus nephritis | 52 weeks
Change in FACIT-F (Functional Assessment of Chronic Illness Therapy-Fatigue)score from baseline | 52 weeks
  FACIT-F scale ranges from 0 to 52 score,and the higher scores indicate a better condition of the subject and less fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: bicheng Liu, Principal Investigator — Institute of Nephrology, Zhong Da Hospital, Southeast University School of Medicine
Locations (1):
- Institute of Nephrology, Zhong Da Hospital, Southeast University School of Medicine, Nanjing, Jiangsu, China